CLINICAL TRIAL: NCT04196062
Title: Prospective, Single Arm Study to Assess the Safety and Performance of the EndoMaster EASE System for the Treatment of Colorectal Lesions
Brief Title: EndoMaster EASE System for Treatment of Colorectal Lesions
Acronym: MASTERCESD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Philip Wai Yan CHIU, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE Ref. No. 2019.331
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Colonic Neoplasms
Keywords: Colonic ESD; Robotic Endoscope
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, Single-Arm Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic ESD (Experimental): Treatment of early colorectal neoplasia / lateral spreading tumors by ESD using EndoMASTER EASE robotic system
  Interventions: Device: EndoMASTER EASE Robotic system for ESD

INTERVENTIONS:
Device: EndoMASTER EASE Robotic system for ESD — EndoMaster EASE System, is a robotic-assisted endoscopy system indicated for endoscopic visualization and therapeutic access to the adult gastrointestinal (GI) tract for endoscopic surgery

SUMMARY:
This is a prospective, single arm study to assess the safety and performance of the EndoMaster EASE (Endoluminal Access Surgical Efficacy) System for the treatment of patients with colorectal neoplasms.

DETAILED DESCRIPTION:
Prospective, single arm study to assess the safety and performance of robotically assisted ESD of superficial colorectal lesions, that otherwise cannot be optimally and radically removed by snare-based techniques

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 85;
2. Suspected intramucosal neoplasm of the colon or rectum, including adenocarcinoma and tubular, tubulovillous, or villous adenomas.

Exclusion Criteria:

1. Informed consent not available;
2. Carcinoma of colon or rectum with known involvement beyond the submucosa;
3. Evidence of distant spread of colon cancer;
4. Presence of another active malignancy;
5. Pregnancy;
6. Patients considered unfit for general anaesthesia;
7. The endoscopic platform cannot reach the target site;
8. Current participation in another clinical research study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Complete (R0) resection | 30 days
  rate of complete (R0) resection defined as en bloc, one-piece resection with histologically confirmed tumour-free lateral and vertical margins

SECONDARY OUTCOMES:
Bleeding during or after the procedure | 30 days
  Bleeding as evidence by
  1. Active bleeding during the robotic ESD procedure
  2. Bleeding after ESD with clinical evidence of 1. Fresh hematemesis; 2. Passage of tarry stool with pulse > 100 or systolic blood pressure < 100; 3. Drop in hemoglobin level of > 4 g/dl
Perforation | 30 days
  Perforation at the ESD site as assessed by endoscopy
Adjunctive procedures to control bleeding | 1 day
  Use of coagrapser / clips
All cause mortality | 30 days
  Mortality
Infection | 30 days
  Clinical sepsis with changes in inflammatory markers as evidence by
  1. clinical symptoms of fever, pulse > 100
  2. radiological evidence of intraperitoneal collection
  3. elevated WBC count of > 10.0
Impairment of renal function | 30 days
  renal failure as evidence of derangement of renal function with elevated creatinin level > 100 mmol/l
Serious Adverse Events | 30 days
  Serous Adverse Events at preocedure and through discharge
Duration of procedure | 1 day
  OT time
Operator assessment of device performance | 1 day
  Operator assessment
Device deficiencies | 1 day
  Device malfunction and Use errors during the ESD procedure as evidence by
  1. cessation of the function of the EndoMASTER EASE system
  2. need to use of the immediate cessation button for the EndoMASTER EASE system
Length of Hospital stay | 30 days
  Length of Hospital Stay
Histology of resected specimen | 30 days
  En bloc resection rate / R0 rate / positive vertical margin / positive lateral margin
Colonoscopy followup | 6 months, 18 months to 3 years
  Healing of operative site / presence of suspicious tissue for biopsy / presence of stricture
Cancer status by cross-sectional imaging (MRI / CT) | 12 months and 3 years
  local recurrence / recurrence at different site in colon / metastatic disease and location
Technical Success | 30 days
  en bloc, one-piece excision of the neoplasm irrespective of histopathology, in the absence of device-related SAE through 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chiu, MD, Study Director — Chinese University of Hong Kong
Locations (1):
- Combined Endoscopy Center, Prince of Wales Hospital, Hong Kong, Hong Kong